CLINICAL TRIAL: NCT06595290
Title: Vietnamese Rapid Acceleration Protocol for Intensifying Drug Therapy in Heart Failure With Reduced Ejection Fraction
Acronym: VN-RAPID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Collaborators: Momentum Research, Inc. (Industry); INSERM UMR-942, Paris, France (Other); University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Vu Hoang Vu, Head of Interventional Cardiology Department, PhD MD, University Medical Center Ho Chi Minh City (UMC)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DHYD-VNRAPID
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Acute Heart Failure (AHF); Acute Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF; STRONG-HF; Acute heart failure; Rapid uptitration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Patients will be managed by their cardiologist according to their usual practice. Follow-up appointments will be scheduled as per the cardiologist's instructions. Participants will return to the recruiting study site for clinical outcome assessment by study investigators at 90 and 180 days post-discharge.
  Interventions: Other: Usual care
- High intensity care (Experimental): This arm follows a structured algorithm for initiating and uptitrating all four pillars of HFrEF oral medications post-randomization (pre-discharge) and during at least 4 visits over 6 weeks post-discharge.
  Interventions: Other: High intensity care

INTERVENTIONS:
Other: High intensity care — This arm follows a structured algorithm for initiating and uptitrating all four pillars of HFrEF oral medications post-randomization (pre-discharge) and during at least 4 visits over 6 weeks post-discharge.
  Arms: High intensity care
Other: Usual care — Patients will be managed by their cardiologist according to their usual practice. Follow-up appointments will be scheduled as per the cardiologist's instructions. Participants will return to the recruiting study site for clinical outcome assessment by study investigators at 90 and 180 days post-discharge.
  Arms: Usual care

SUMMARY:
VN-RAPID is an open-label, multicenter, randomized controlled trial evaluating the safety and efficacy of in-hospital initiation and rapid up-titration of four-pillar therapy for hospitalized Asian patients with acute heart failure (AHF) and reduced ejection fraction (HFrEF). The study compares a standardized protocol of intensified treatment (high-intensity care arm) with usual care in patients with elevated NT-proBNP levels who are not on optimal HFrEF medications. The high-intensity care arm involves initiation of all four pillars of HFrEF therapy (RAS inhibitor, beta-blocker, MRA, and SGLT2i) before discharge, followed by a structured 6-week outpatient up-titration process with frequent follow-ups. The study aims for 75% of target doses for RAS inhibitors and beta-blockers, considering the lower blood pressure tendency in Asian populations. Participants will be followed for 180 days to assess clinical outcomes.

DETAILED DESCRIPTION:
VN-RAPID is an open-labeled, multicenter, randomized study modeled after the STRONG-HF trial with the aim to evaluate the safety and efficacy of a standardized protocol of in-hospital initiation and rapid up-titration of all four pillars therapy for hospitalized acute heart failure (AHF) Asian patients with reduced ejection fraction (HFrEF). The study will enroll patients hospitalized with AHF with elevated NT-proBNP levels and not receiving optimal doses of oral HFrEF medications within 48 hours of discharge and are hemodynamically stable. These participants will be randomized in a 1:1 ratio to either usual care (named "usual care" arm) or intensification of treatment with all four pillars including RAS inhibitor (either ACEi or ARB or ARNi), beta-blocker, MRA and SGLT2i (named "high intensity care" arm). In the latter arm, the patients will be prescribed all four pillars before discharge with at least ¼ target dose. To ensure patient safety during the outpatient uptitration process, the high intensity care group will undergo thorough assessments at four follow-up appointments over a six-week period post-discharge, including physical examinations for signs and symptoms of congestion, laboratory tests such as NT-proBNP, serum creatinine, electrolytes. In consideration of the generally lower blood pressure observed in Asian populations, VN-RAPID establishes a target dose for RAS inhibitors and beta-blockers at 75% of the conventional target dose during outpatient uptitration. All participants will be followed through 180 days from randomization with 2 additional visits at 90-day and 180-day to assess clinical endpoints.

Primary objective:

To demonstrate that the VN-RAPID protocol-comprising in-hospital initiation and rapid outpatient uptitration of HFrEF four-pillar medical therapy, with lower target doses (75% of conventional) for RAS inhibitors and beta-blockers-is superior to usual care in reducing 180-day all-cause mortality or heart failure rehospitalization among Vietnamese patients hospitalized with acute heart failure and reduced ejection fraction.

Secondary objectives:

* To demonstrate the superiority of the VN-RAPID protocol, compared to usual HFrEF care, in reducing 180-day all-cause mortality
* To demonstrate the superiority of the VN-RAPID protocol, compared to usual HFrEF care, in reducing 180-day heart failure rehospitalization
* To demonstrate the superiority of the VN-RAPID protocol, compared to usual HFrEF care, in reducing 90-day all-cause mortality or heart failure rehospitalization
* To demonstrate the superiority of the VN-RAPID protocol, compared to usual HFrEF care, in reducing left ventricular remodeling by evaluation of LVEDV, LVEF on echocardiography at 90-day and 180-day
* To demonstrate the superiority of the VN-RAPID protocol, compared to usual HFrEF care, in reducing 90-day and 180-day congestion index score
* To evaluate the safety and tolerability of the VN-RAPID protocol

ELIGIBILITY:
Inclusion Criteria:

1. Hospital admission with diagnosis of acute heart failure assessed by clinical signs and symptoms of congestion and radiographic, biological tests (if admitted with acute coronary syndrome, required at least Killip class II or clear evidence of congestion on admission assessed by chest x-ray or lung ultrasound and/or pulmonary congestion requiring intravenous treatment)
2. Female or male patients ≥ 18 years old
3. At randomization:

   1. Systolic blood pressure > 90 mmHg (at least 2 measurements on 2 different occasions) and
   2. Heart rate ≥ 60 bpm (at least 2 measurements on 2 different occasions) and
   3. Serum potassium ≤ 5.0 mmol/L
4. Left ventricular ejection fraction (LVEF) ≤ 40% assessed locally by Simpson's Biplane method via echocardiography (if multiple LVEF measurements, the last one performed prior to randomization should be considered as the qualifying measurement)
5. Persistent congestion at the time of randomization with pre-discharge NT-proBNP ≥ 1500 ng/L
6. HFrEF medications at randomization:

   1. ≤ ¼ RASi/ARNi target dose and
   2. ≤ ¼ beta-blocker target dose and
   3. ≤ ½ MRA dose
7. Obtained written informed consent form

Exclusion Criteria:

1. Clearly documented intolerance to high doses of RASi/ARNi or beta-blockers
2. Absolute contraindication to usage of RASi/ARNi or beta-blocker or MRA or SGLT2i as per ESC 2021/ACC 2022 Heart failure guideline
3. LVEF >40% assessed by echocardiography on the latest measurement prior to discharge
4. Renal disease or eGFR < 30 mL/min/1.73m2 (as estimated by the CKD-EPI 2021 or the simplified MDRD) at Screening or history of dialysis.
5. Significant pulmonary disease contributing substantially to the patients' dyspnea such as FEV1< 1 liter or need for chronic systemic or nonsystemic steroid therapy, or any kind of primary right heart failure such as primary pulmonary hypertension or recurrent pulmonary embolism.
6. Implantation of cardiac resynchronization device or underwent coronary artery bypass graft surgery within 3 months
7. Myocardial infarction, unstable angina or cardiac surgery within 3 months, or cardiac resynchronization therapy (CRT) device implantation within 3 months, or percutaneous coronary intervention (PCI), within 1 month prior to Screening.
8. AHF triggered primarily by a correctable etiology such as significant arrhythmia (e.g., sustained ventricular tachycardia, or atrial fibrillation/flutter with sustained ventricular response >130 beats per minute, or bradycardia with sustained ventricular arrhythmia <45 beats per minute), infection, severe anemia, pulmonary embolism, exacerbation of COPD, planned admission for device implantation or severe non-adherence leading to very significant fluid accumulation prior to admission and brisk diuresis after admission. Troponin elevations without other evidence of an acute coronary syndrome are not an exclusion.
9. Uncorrected thyroid disease, active myocarditis, or known amyloid or hypertrophic obstructive cardiomyopathy.
10. History of heart transplant or on a transplant list, or using or planned to be implanted with a ventricular assist device.
11. Sustained ventricular arrhythmia with syncopal episodes within the 3 months prior to screening that is untreated.
12. Presence at Screening of any hemodynamically significant valvular stenosis or regurgitation, except mitral or tricuspid regurgitation secondary to left ventricular dilatation, or the presence of any hemodynamically significant obstructive lesion of the left ventricular outflow tract.
13. Active infection at any time during the AHF hospitalization prior to Randomization based on abnormal temperature and elevated WBC or need for intravenous antibiotics.
14. Stroke or TIA within the 3 months prior to Screening.
15. Primary liver disease considered to be life threatening.
16. Psychiatric or neurological disorder, cirrhosis, or active malignancy leading to a life expectancy < 6 months.
17. Prior (defined as less than 30 days from screening) or current enrollment in a CHF trial or participation in an investigational drug or device study within the 30 days prior to screening
18. Discharge for the AHF hospitalization anticipated to be > 14 days from admission, or to a long-term care facility. Randomization must occur within 12 days following admission and at within 2 days prior to anticipated discharge.
19. Inability to comply with all study requirements, due to major comorbidities, social or financial issues, or a history of noncompliance with medical regimens, that might compromise the patient's ability to understand and/or comply with the protocol instructions or follow-up procedures
20. Pregnant or nursing (lactating) women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
180-day all-cause death or heart failure rehospitalization | 180 days post-discharge
  Cumulative risk of either rehospitalization for heart failure or death at 180 days

SECONDARY OUTCOMES:
90-day all-cause mortality or heart failure rehospitalization | 90 days post-discharge
  Cumulative risk of either rehospitalization for heart failure or death at 90 days
180-day all-cause mortality | 180 days post discharge
  Cumulative risk of death at 180 days
180-day heart failure rehospitalization | 180 days post discharge
  Cumulative risk of heart failure rehospitalization at 180 days
Change in NT-proBNP at 180-day | 180 days post-discharge
  Change of NT-proBNP levels from pre-discharge to 180 days post-discharge
Change in left ventricular end-diastolic volume at 180-day | 180 days post discharge
  Change of left ventricular end-diastolic volume (LVEDV) from pre-discharge to 180 days post-discharge. LVEDV is measured in mL on echocardiography.
Change in left ventricular ejection fraction at 180-day | 180 days post discharge
  Change of left ventricular ejection fraction (LVEF) from pre-discharge to 180 days post-discharge. LVEF is measured in % on echocardiography using Simpson biplane method.

OTHER OUTCOMES:
Change in congestion score at 180-day | 180 days post discharge
  Change of congestion score from pre discharge to 180 days post discharge. The congestion score was calculated as a sum of points gained for:
  * Presence (1 point)/absence (0 points) of edema
  * Presence (1 point)/absence (0 points) of pulmonary rales
  * JVP lower than 6 cm (0 points)/equal to or greater than 6 cm (1 point) A congestion score of 0 was deﬁned as a criterion for successful decongestion.
Change on lung ultrasound at 180-day | 180 days post discharge
  Change of the number of B lines measured at pre discharge to 180 days post discharge. B lines are measured on lung ultrasound using a 4-zone scanning protocol. 0 B line indicates no congestion.

CONTACTS AND LOCATIONS:
Locations (4):
- Vietnam (4):
  - An Giang Heart Hospital, Long Xuyen, An Giang
  - Thong Nhat Hospital, Ho Chi Minh City, Ho Chi Minh City
  - University Medical Center Ho Chi Minh City, Ho Chi Minh City, Ho Chi Minh City
  - Quang Tri Province Hospital, Đông Hà, Quang Tri

IPD SHARING:
Plan to Share IPD: No